CLINICAL TRIAL: NCT07319143
Title: Utilizing Transcranial Direct Current Stimulation (tDCS) to Alleviate Subthreshold Depression Via Distinct Positive and Negative Emotion Pathways
Brief Title: The Effect of Transcranial Direct Current Stimulation (tDCS) in Improving Emotion Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Zhengxi Shao, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA240670; 17600425 (Other Grant/Funding Number: Research Grants Council)
Record Dates: First submitted 2025-12-06; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Subthreshold Depression; Positive Emotions; Negative Emotions; Anhedonia
Keywords: Transcranial Direct Current Stimulation; Subthreshold Depression; Emotion; Neuromodulation
MeSH Terms: conditions — Anhedonia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IDLPFC (Experimental): This intervention is a 20 minutes per session, two-week tDCS neuromodulation of IDLPFC region (anode: F3, cathode: FP2) designed to reduce depressive symptoms via enhancing positive emotion functions, thereby reducing anhedonia.
  Interventions: Device: Transcranial Direct Current Stimulation
- rVLPFC (Experimental): This intervention is a 20 minutes per session, two-week tDCS neuromodulation of rVLPFC region (anode: F6, cathode: FP1) designed to reduce depressive symptoms via regulating negative emotion functions, thereby reducing depressed mood.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham (Sham Comparator): This is a 20 minutes per session, two-week Sham comparator of IDLPFC/rVLPFC region, participants will receive tDCS for 90 seconds at either IDLPFC/rVLPFC at the beginning of each session to stimulate real neuromodulation.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — TDCS is a non-invasive, safe, inexpensive, convenient and effective method to modulate brain and emotion functions. During tDCS, a mild electric current is passed between the anodal and cathodal electrodes on the scalp, which respectively excites and inhibits local and downstream neuronal activity, as well as modulating interregional connectivity strength. Compared to other neurostimulation methods such as Transcranial Magnetic Stimulation, tDCS side effects tend to be milder and transient, even if being administered for multiple sessions, making it suitable to be widely applied on clinical and subclinical populations.
  Other Names: tDCS

SUMMARY:
The goal of this clinical trial is to investigate how transcranial direct current stimulation (tDCS) affects emotion functions in young adults aged 18-35 from the local community, including both male and female participants. The main question[s] it aims to answer are:

* Does tDCS improve emotional functions, such as mood regulation and motivation, in individuals with subthreshold depression (StD)?
* Can tDCS enhance emotional regulation compared to a sham stimulation (placebo)?

Researchers will compare participants receiving tDCS on either the left dorsolateral prefrontal cortex (lDLPFC) or right ventrolateral prefrontal cortex (rVLPFC) with those receiving sham stimulation to see if tDCS has a stronger effect on emotional functions.

Participants will:

* Complete online and in-person screening to assess depressive symptoms using the Chinese version of the Beck Depression Inventory II (C-BDI-II) and be selected based on their depressive symptoms (C-BDI-II score ≥ 13).
* Be randomly assigned to one of three groups: lDLPFC tDCS, rVLPFC tDCS, or Sham control group (1:1:1 ratio).
* Receive 10 sessions of tDCS or Sham tDCS over 2 weeks, with each session lasting 20 minutes.
* Complete assessments at baseline, post-intervention, 1-month follow-up, and 3-month follow-up, with each assessment lasting 2-2.5 hours. This includes questionnaires and perform emotional and cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Fluency in Cantonese or Mandarin
* Normal or corrected-to-normal vision and hearing
* IQ > 75% Quantile in Raven's SPM
* At least 9 years of formal education
* Right-handedness

Exclusion Criteria:

* Past or current major physical illness or psychiatric disorders
* Use of psychotropic medication in the past 6 months
* Pregnancy (for women)
* Any condition that prevents safe tDCS use (e.g., brain injury, implants)
* Previous participation in neuromodulation in the past 3 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Beck Depression Inventory-II Chinese Version measures change in depressive symptoms. The total score range is 0-63, higher score indicates more severe depressive symptoms.

SECONDARY OUTCOMES:
Affective trait | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Chinese Affect Scale measures changes in positive and negative affective traits. Both the positive affect and the negative affect subscales have a score range of 0-40, with higher scores indicating higher levels of positive affect trait and negative affect trait respectively.
Anhedonia severity | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The dimensional anhedonia rating scale measures change in anhedonia severity on distinct physical/social domain. The scale comprises four subscales: Hobbies (4 items; score range 0-16), Food/Drink (4 items; score range 0-16), Social Activities (4 items; score range 0-16), and Sensory Experience (5 items; score range 0-20), with higher scores on each subscale indicating less anhedonia severity within the corresponding domain.
Anhedonia symptoms | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Chapman Physical/Social Anhedonia scales assess change in anhedonia symptoms in physical and social domains. The Chapman Physical Anhedonia Scale consists of 61 true-false items with a total score range of 0-61, and the Chapman Social Anhedonia Scale consists of 40 true-false items with a total score range of 0-40. For both scales, higher scores indicate higher levels of anhedonia.
Behavioural motivation trait | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Behavioural Activation and Inhibition Scale measures change in reward-driven approaching and punishment-driven avoidance tendencies. The Behavioural Inhibition System scale consists of 7 items with a score range of 7-28, with higher scores indicating higher behavioural inhibition. The Behavioural Activation System scale comprises three subscales: Drive (4 items; score range 4-16), Fun Seeking (4 items; score range 4-16), and Reward Responsiveness (5 items; score range 5-20). Higher scores on each BAS subscale indicate higher levels of behavioural activation within the corresponding domain.
Emotion regulation function | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Cognitive Emotion Regulation Questionnaire measures change in emotion regulation functions. The scale comprises nine subscales, Self-Blame, Acceptance, Rumination, Positive Refocusing, Refocus on Planning, Positive Reappraisal, Putting into Perspective, Catastrophising, and Other-Blame. Each consisting of 2 items with a score range of 2-10. Higher scores on each subscale indicate greater habitual use of emotion regulation strategy.
Coping to adversity | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Brief Coping Orientation to Problems Experienced inventory measures change in people's coping strategies to hardships. The problem-focused subscale consist of 8 items (score range 4-32). The emotion-focused subscale consists of 12 items (score range 4-46). The avoidant/dysfunctional coping subscale consists of 8 items (score range 4-32). In each subscale, higher scores indicate greater use of the corresponding coping strategy.
Reward sensitivity | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Temporal Experience of Pleasure Scale assesses change in sensitivity towards both anticipatory and consummatory pleasurable experience. The scale comprises four subscales: Abstract Anticipatory Pleasure (4 items; score range 4-24), Contextual Anticipatory Pleasure (5 items; score range 5-30), Abstract Consummatory Pleasure (6 items; score range 6-36), and Contextual Consummatory Pleasure (4 items; score range 4-24), with higher scores on each subscale indicating greater capacity to experience pleasure from reward.
Apathy symptom | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Apathy Evaluation Scale-Self measures change in emotional indifference and apathy (lack of motivation). The scale consists of 18 items, yielding a total score range of 0-54, with higher scores indicating greater emotional indifference and higher levels of apathy.
Perceived loneliness | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The brief UCLA Loneliness Scale measures change in the participants' subjective loneliness. The scale consists of 6 items yielding a total score range of 6-24, with higher scores indicating higher levels of perceived loneliness.
Stress level | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The 10-item Perceived Stress Scale measures change in perceived stressful experiences. The scale consists of 10 items yielding a total score range of 0-40, with higher scores indicating higher levels of perceived stress.
Emotion ratings of words | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Emotion Rating Task measures changes in participants' feeling and motivation to positive social, positive non-social, negative social and negative non-social word stimuli.
Instrumental behavioural motivation | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Monetary Incentive Delay task measures change in behavioural motivations to obtain rewards or to avoid punishment.
Emotional inhibition control | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The Emotion Stroop task measures change in participants' inhibition control of emotional processing.
Cognitive control function | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The colour stroop measures change in cognitive control and inhibition functions.
Working memory | Baseline (Day 1), Post-Intervention (Day 15), 1-Month Follow-up (Day 45), 3-Month Follow-up (Day 105)
  The N-back task measures change in the participants' working memory capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No